CLINICAL TRIAL: NCT03588923
Title: A Randomized, Double-blind, Placebo-controlled Phase I Study to Assess Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of SH229 in Patients With Hepatitis C Virus (HCV) Infection
Brief Title: Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of SH229 in Patients With HCV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHC005-I-03
Record Dates: First submitted 2018-07-02; First posted 2018-07-17 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: HCV Infection
Keywords: HCV; NS5B; SH229
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): SH229 (400 mg) or matching placebo, once daily
  Interventions: Drug: SH229; Drug: Placebos
- Cohort 2 (Active Comparator): SH229 (600 mg) or matching placebo, once daily
  Interventions: Drug: SH229; Drug: Placebos
- Cohort 3 (Active Comparator): SH229 (800 mg) or matching placebo, once daily
  Interventions: Drug: SH229; Drug: Placebos

INTERVENTIONS:
Drug: SH229 — tablet, oral, 400 mg once daily for 3 days
  Arms: Cohort 1
Drug: Placebos — tablet, oral, once daily for 3 days
  Arms: Cohort 1
Drug: SH229 — tablet, oral, 600 mg once daily for 3 days
  Arms: Cohort 2
Drug: Placebos — tablet, oral, once daily for 3 days
  Arms: Cohort 2
Drug: SH229 — tablet, oral, 800 mg once daily for 3 days
  Arms: Cohort 3
Drug: Placebos — tablet, oral, once daily for 3 days
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and antiviral activity of single and multiple ascending doses of SH229 in patients with chronic hepatitis C Virus infection.

DETAILED DESCRIPTION:
A total of 30 evaluable patients will be enrolled in this study. The planned dose levels are 400, 600, and 800 mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are willing to voluntarily take effective contraceptive measures from screening to 6 months after the last dose;
* 18-65 years of age;
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive, and a body weight ≥50 kg for males and ≥45 kg for females;
* No previous treatment with any direct-acting antiviral (DAA) drugs for HCV, such as Boceprevir, Telaprevir, Simeprevir, Sofosbuvir, Daclatasvir, Asunaprevir;
* No antiviral treatment such as immune modulators, thymosin or other immune stimulating factors, interferon, or Chinese herbs in the past 6 months;
* HCV RNA ≥10*5 IU/mL at screening (Roche COBAS Taqman);
* Chronic genotype 1-6 HCV Infection;
* Serum ALT ≤10 times ULN;
* FibroScan score ≤17.5kPa within 6 months before screening or at screening, or absence of cirrhosis within 12 months before screening;
* Subjects are capable of understanding and complying with the protocol and have signed the informed consent form.

Exclusion Criteria:

* Smoke more than 5 cigarettes per day within three months prior to screening;
* Subjects allergic to the study drug (including its excipients) or subjects who are prone to allergies;
* History of drug and/or alcohol abuse (alcohol consumption exceeding 14 units per week: 1 unit = 285 mL of beer, or 25 mL of hard liquor, or 100 mL of wine);
* Blood donation or massive blood loss (> 450 mL) within three months prior to screening;
* History of any non-HCV liver diseases, including but not limited to hemochromatosis, primary biliary cirrhosis, Wilson's disease, autoimmune hepatitis, drug or alcoholic hepatitis, non-alcoholic steatohepatitis, etc.;
* Subjects with dysphagia or with any gastrointestinal disorders (or postoperative conditions) that may affect the study drug absorption;
* Subjects with any diseases that increase the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
* Use of any drugs that alter liver enzyme activity within 28 days prior to screening;
* Use of any prescription drugs, over-the-counter drugs, vitamin products or herbal medicines within 14 days prior to screening;
* Use of special diet (including dragon fruit, mango, grapefruit, etc.), strenuous activities or other factors that may affect the disposition of the study drug within 2 weeks prior to screening;
* Concomitant use of strong inhibitors or inducers of CYP3A4, P-gp or Bcrp, such as itraconazole, ketoconazole or dronedarone;
* Subjects with major changes in diet or exercise habits recently;
* Participation in other clinical trials within three months prior to enrollment;
* Electrocardiogram abnormalities with clinical significance;
* Laboratory tests with clinical significance or other clinical findings that indicate clinically significant diseases not associated with HCV infection (including but not limited to gastrointestinal, renal, hepatic, neurologic, hematological, endocrine, pulmonary, psychiatric, cardiovascular diseases);
* Pregnant or lactating women;
* Creatinine clearance ≤ 60 mL/min;
* Evidence of co-infection with HBV, HIV, or syphilis;
* Child-Pugh Grade B or C;
* Clinically significant hepatic decompensation including but not limited to, hepatic encephalopathy, hepatocellular carcinoma, variceal bleeding, ascites, etc.;
* Use of chocolate, food or beverages containing caffeine or xanthine within 24 hours prior to dosing;
* Use of products containing alcohol within 24 hours prior to dosing;
* Subjects with urine drug screening test positive, or with history of drug abuse in the past 5 years;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to Day 10
Antiviral effects of SH229, as measured by HCV RNA levels | up to Day 10

SECONDARY OUTCOMES:
Time to peak plasma concentration(Tmax) | up to Day 10
Peak plasma concentration(Cmax) | up to Day 10
Half-life time(t1/2) | up to Day 10
Area under the plasma concentration versus time curve(AUC) | up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — Phase I Clinical Trial Unit, The First Hospital of Jilin University
Locations (1):
- Phase I Clinical Trial Unit, The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No